CLINICAL TRIAL: NCT05040230
Title: EEG Encephalopathy Patterns in Immune Effectors Cells-associated Neurotoxicity Syndrome : a Prospective Observational Study
Brief Title: EEG Encephalopathy Patterns in Immune Effectors Cells-associated Neurotoxicity Syndrome (ICANS)Lay Language
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0287
Record Dates: First submitted 2021-06-02; First posted 2021-09-10 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Immune Effector Cell Encephalopathy; Neurotoxicity
MeSH Terms: conditions — Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Immune effectors cells-associated neurotoxicity syndrome (ICANS) is one of the most clearly defined acute toxicities after CAR-T cells infusion.

The investigators conducted a prospective cohort study of all patients who received CAR T cell infusions on the hematology department from Montpellier University Medical Center.

Each patient was assessed between the 6th and 8th day after infusion by a neurological clinical examination, an electroencephalogram, and a brain MRI.

The aim of the studies is to describe the EEG pattern associated with ICANS.

DETAILED DESCRIPTION:
The investigators will conduct a prospective cohort study of all patients who received CAR T cell infusions in the hematology department from Montpellier University Medical Center. To be eligible for enrollment, patients should have to be 18 years of age or older. All the patients will have histologically confirmed: diffuse large B-cell lymphoma, B-cell acute lymphoblastic leukemia, follicular lymphoma, or mantle cell lymphoma.

Each patient will have a PET CT before infusion to determine metabolic response status according to the LUGANO grading classification. All patients will have preconditioning brain imaging by MRI.

Each patient will be assessed between the 6th and 8th day after infusion by a neurological clinical examination, an electroencephalogram, and a brain MRI.

Patients will be called back one month later to report any new neurological event and an EEG was performed if abnormalities were found on the first.

All neurological symptoms documented in daily progress notes will be catalogued. The investigators will use ASTCT ICANS Consensus Grading for Adults to evaluate neurotoxicity.

ELIGIBILITY:
Inclusion criteria:

* histologically confirmed: diffuse large B-cell lymphoma, B-cell acute lymphoblastic leukemia, follicular lymphoma, or mantle cell lymphoma.
* with infusion of CAR T-cells

Exclusion criteria:

- Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: a prospective cohort study of all patients who received CAR T cell infusions on the hematology department from Montpellier University Medical Center between September 2020 and July 2021
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
to assess the sensitivity of EEG for diagnosis of ICANS. | day 1
  bandwidth of the EEG which will be assessed during the period of study :
  1. background frequencies : alpha, theta or delta
  2. reactivity on opening the eyes : yes or not
  3. organization of background activity : present or absent
  4. presence of paroxysmal activities : yes or not

SECONDARY OUTCOMES:
to identify a biomarker for ICANS | day 1
  to identify a biomarker for ICANS

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Ayrignac, MD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC